CLINICAL TRIAL: NCT03448991
Title: Effect of NPO Time and Type of Food Intake on Preoperative Residual Gastric Content and pH
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Patcharee Sriswasdi, Principal investigator, Boston Children's Hospital
Other Study IDs: IRB-P00027981
Record Dates: First submitted 2018-02-20; First posted 2018-02-28 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Fasting; Pediatric ALL
Keywords: NPO time; Gastric content; Gastric pH
MeSH Terms: conditions — Fasting; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to normal physiology, the longer fasting period allows food particles to pass stomach through small intestines to minimize intragastric content. The practice guidelines recommend 2-hour fasting period for clear fluid (including water, pulp-free juice and tea or coffee without milk), 4- hour fasting period for breast milk and 6-hour fasting period for non-human milk and solid food to reduce risks of pulmonary aspiration. As a result of longer fasting period, patients tend to experience preoperative dehydrated states and intraoperative hypotension. Patients' demographic data will be obtained from charts. Parents will be asked for type, volume of fluid/food intake and NPO time.

This study will be done at BCH's Gastroenterology Procedure Unit (GPU) theaters to measure actual intragastric volume and pH at the beginning esopagogastroduodenoscopy procedures. We hope to demonstrate the relationship between NPO time and actual intragastric volume which provide sufficient data of NPO time to ensure patient's safety.

DETAILED DESCRIPTION:
This study is a prospective observational cohort study which will be conducted in 2 parts including preoperative and intraoperative periods.

* Preoperative period, patients' demographic information will be collected along with NPO history including times, type ,amount of preoperative fluid/ food intake and patients' anxiety score.
* Intraoperatively, at the beginning of EGD procedure, total volume of intragastric content(ml) and gastric acidity will be measured.

We plan to offer participation to all patients or parents of patients' ages 0-17 years who are scheduled for EGD at GPU, BCH Longwood campus and are fluent in English. A brochure describing our study in English will be given to patients or their families on the day of surgery. If the patient or family agrees to participate in this study, the study will be provided in the GPU theaters.

ELIGIBILITY:
Inclusion Criteria:

- All patients who aged 0-17 years scheduled for EGD procedure.

Exclusion Criteria:

- Patients who required emergency EGD procedures and patients with active upper GI bleeding.

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will include all patients who aged 0-17 years scheduled for EGD procedure at GPU, Boston Children's Hospital, Longwood.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Actual intragastric content volume (ml) | 1 day
  Actual intragastric content volume (ml) which is suctioned from each pediatric patient is measured

SECONDARY OUTCOMES:
Correlation between NPO time(hr) and intraoperative intragastric content volume(ml). | 1 day
  Correlation between NPO time(hr) and intraoperative intragastric content volume(ml).
Correlation between NPO time(hr) and intraoperative intragastric content acidity (pH). | 1 day
  Correlation between NPO time(hr) and intraoperative intragastric content acidity (pH).
Incidence of perioperative hypotension | 1 day
  Hypotension is defined as 20% reduction of normal systolic blood pressure for any age groups
Incidence of pulmonary aspiration risk. | 1 day
  Pulmonary aspiration is defined by the regurgitation of gastric contents into the larynx and the respiratory tract and cause a syndrome of progressive dyspnea, hypoxia, bronchial wheeze and patchy collapse, consolidation on chest X-ray or all.
Correlation between preoperative patient's anxiety score and actual intragastric content volume (ml) | 1 day
  Correlation between preoperative patient's anxiety score and actual intragastric content volume (ml)
Incidence of surgery delay or cancellation due to NPO guideline violation | 1 day
  Surgery delay is defined when the patient's queue is postponed in order to wait for proper NPO time
Actual pH of intragastric content | 1 day
  Actual pH of intragastric content which is suctioned from each pediatric patient is measured

CONTACTS AND LOCATIONS:
Overall Officials: Patcharee Sriswasdi, MD., Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston children hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration: Application to Healthy Patients Undergoing Elective Procedures: An Updated Report by the American Society of Anesthesiologists Task Force on Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration. Anesthesiology. 2017 Mar;126(3):376-393. doi: 10.1097/ALN.0000000000001452. No abstract available. PMID 28045707
- [Result] Smith I, Kranke P, Murat I, Smith A, O'Sullivan G, Soreide E, Spies C, in't Veld B; European Society of Anaesthesiology. Perioperative fasting in adults and children: guidelines from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2011 Aug;28(8):556-69. doi: 10.1097/EJA.0b013e3283495ba1. PMID 21712716
- [Result] Maltby JR, Sutherland AD, Sale JP, Shaffer EA. Preoperative oral fluids: is a five-hour fast justified prior to elective surgery? Anesth Analg. 1986 Nov;65(11):1112-6. PMID 3767008
- [Result] Andersson H, Zaren B, Frykholm P. Low incidence of pulmonary aspiration in children allowed intake of clear fluids until called to the operating suite. Paediatr Anaesth. 2015 Aug;25(8):770-777. doi: 10.1111/pan.12667. Epub 2015 May 4. PMID 25940831
- [Result] Phillips S, Daborn AK, Hatch DJ. Preoperative fasting for paediatric anaesthesia. Br J Anaesth. 1994 Oct;73(4):529-36. doi: 10.1093/bja/73.4.529. PMID 7999497
- [Result] Dennhardt N, Beck C, Huber D, Sander B, Boehne M, Boethig D, Leffler A, Sumpelmann R. Optimized preoperative fasting times decrease ketone body concentration and stabilize mean arterial blood pressure during induction of anesthesia in children younger than 36 months: a prospective observational cohort study. Paediatr Anaesth. 2016 Aug;26(8):838-43. doi: 10.1111/pan.12943. Epub 2016 Jun 13. PMID 27291355
- [Result] Song IK, Kim HJ, Lee JH, Kim EH, Kim JT, Kim HS. Ultrasound assessment of gastric volume in children after drinking carbohydrate-containing fluids. Br J Anaesth. 2016 Apr;116(4):513-7. doi: 10.1093/bja/aew031. PMID 26994229
- [Result] Schmitz A, Kellenberger CJ, Liamlahi R, Studhalter M, Weiss M. Gastric emptying after overnight fasting and clear fluid intake: a prospective investigation using serial magnetic resonance imaging in healthy children. Br J Anaesth. 2011 Sep;107(3):425-9. doi: 10.1093/bja/aer167. Epub 2011 Jun 14. PMID 21676893